CLINICAL TRIAL: NCT00388245
Title: Myocardial Revascularization in Patients With Ischemic Cardiomyopathy: a Comparison Between Percutaneous Coronary Intervention and Coronary Artery Bypass Surgery
Brief Title: Revascularization in Heart Failure Trial - REHEAT 2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Science and Higher Education, Poland (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0213/P01/2006/31
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2006-10-16 (Estimated); Status verified 2006-10

CONDITIONS: Left Ventricular Ejection Fraction; Myocardial Revascularization; Ischemic Heart Disease
Keywords: PCI; CABG; Ejection Fraction; Myocardial Revascularization
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention
Procedure: Coronary Artery Bypass Grafting

SUMMARY:
REHEAT 2 study is designed as a prospective, randomised trial comparing two strategies of myocardial revascularisation (PCI vs CABG) in patients with ischemic cardiomyopathy and low left ventricular ejection fraction.Patients will undergo in random way PCI or CABG procedure. The aim the study is to assess the improvement of left ventricle systolic function and comparing recent (30 days) and late (12 months) results of surgical (CABG) and percutaneous (PCI) revascularization.

DETAILED DESCRIPTION:
Heart failure constitutes one of basic problems of contemporary cardiology. It is most commonly caused by ischaemic heart disease, which as an etiologic factor, has a negative impact on prognosis. On the other hand, decreased left ventricular ejection fraction is the most important prognostic factor in patients with ischaemic heart disease. Annual mortality among patients with ejection fraction below 35% accounts for 17%, and in a group with ejection fraction below 25% reaches 24%. Most of multicenter studies (e.g. ARTS, BARI, ERACI) comparing results of percutaneous and surgical revascularisation in ischemic heart disease pertain to patients with normal or minimally decreased left ventricular ejection fraction, excluding patients with left ventricular ejection fraction lower than 35%. Current medical standards indicate the surgical way as a method of choice in treatment of patients with ischemic cardiomyopathy.

In early nineties the procedures of percutaneous angioplasty in patients with depressed left ventricular function were connected with comparable to CABG risk of death (5-10%).

The intensive progress of percutaneous procedures contributed PCI is competitive method of revasularization to CABG. Our knowledge about the efficacy of above mentioned methods in patients with ischemic heart failure is scarce until now. It was proved, that patients with viable myocardium assessed in dobutamine stress echocardiography or MRI benefit mostly from myocardial revascularization. Repeat revascularization during follow up occurred more frequently in patients after PCI, so that introduction of coronary stents, especially drug eluting stents (DES) could significantly improve the clinical outcome after PCI procedures. The administration of antiplatelet drugs (IIb/IIIa platelet receptor inhibitors) have considerably improved the short and long-term results of PCI so that it is interesting if they could have beneficial effect on clinical outcome of patients with ischemic heart failure. In the field of cardiac surgery the method of left ventricle reconstruction in patients with ischemic cardiomyopathy (STICH Trial) seems to be promising.

Therefore, the comparison of innovative methods of percutaneous and surgical revascularization may influence current medical standards concerning patients with ischemic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic coronary artery disease (angina CCS class 1)
* left ventricle ejection fraction <40%
* coronary artery lesions suitable for percutaneous or surgical myocardial revascularisation
* evidence for viability of the myocardium
* written inform consent for the study

Exclusion Criteria:

* age <18 years
* acute myocardial infarct with ST elevation within 30 days
* concomitant congenital heart disease
* mitral regurgitation required surgical intervention
* history of bleeding diathesis, coagulopathy or abnormal bleeding within the previous 30 days.
* major surgery within the previous 6 weeks
* stroke or transient ischemic attack (TIA) within the previous 6 weeks
* history of hemorrhagic stroke
* uncontrolled hypertension
* chronic renal insufficiency with creatinine >2.0 mg/dl
* platelet count <100.000/mm3
* hematocrit <30%
* PT >1,2 times control
* positive pregnancy test
* any disease that may shorten the life expectancy of the patient
* the patient is currently participating in another research study

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2007-01; Study Completion 2008-12

PRIMARY OUTCOMES:
LV ejection fraction after 1 year since the index procedure

SECONDARY OUTCOMES:
in-hospital and 30 day major adverse events (MAE) and major adverse cardiovascular events (MACE) defined as: death, AMI, stroke, acute heart failure, re-CABG, re-PTCA;
major adverse coronary and cerebrovascular events during 1 year follow-up (MACCE): death, repeat revascularisation, AMI, unstable angina, heart transplantation, heart failure stroke;
long term survival;
severity of angina, exercise and functional capacity along with assessment of quality of life in one year observation.

CONTACTS AND LOCATIONS:
Overall Officials: Pawel E Buszman, Prof, Study Director — 3-rd Division of Cardiology, University School of Silesia, Poland; Michal Tendera, Prof, Study Chair — 3-rd Division of Cardiology, University School of Silesia, Poland; Andrzej Bochenek, Prof, Principal Investigator — 1-st Division of Cardiosurgery, University School of Silesia, Poland; Robert J Gil, Prof, Principal Investigator — Invasive Cardiology Department, Central Clinic Hospital, Warsaw, Poland; Piotr Ponikowski, Prof, Principal Investigator — Heart Disease Department, Military Clinic Hospital, Wroclaw, Poland
Locations (4):
- Poland (4):
  - University School of Silesia, 1-st Department of Cardiosurgery, Katowice, Silesian Voivodeship
  - University School of Silesia, 3-rd Department of Cardiology, Coronary Care Unit, Katowice, Silesian Voivodeship
  - Central Clinic Hospital, Warsaw
  - Military Clinic Hospital, Wroclaw

REFERENCES:
- [Result] Serruys PW, Ong AT, van Herwerden LA, Sousa JE, Jatene A, Bonnier JJ, Schonberger JP, Buller N, Bonser R, Disco C, Backx B, Hugenholtz PG, Firth BG, Unger F. Five-year outcomes after coronary stenting versus bypass surgery for the treatment of multivessel disease: the final analysis of the Arterial Revascularization Therapies Study (ARTS) randomized trial. J Am Coll Cardiol. 2005 Aug 16;46(4):575-81. doi: 10.1016/j.jacc.2004.12.082. PMID 16098418
- [Result] Scholz KH, Dubois-Rande JL, Urban P, Morice MC, Loisance D, Smalling RW, Figulla HR. Clinical experience with the percutaneous hemopump during high-risk coronary angioplasty. Am J Cardiol. 1998 Nov 1;82(9):1107-10, A6. doi: 10.1016/s0002-9149(98)00566-9. PMID 9817489
- [Result] Shawl FA, Quyyumi AA, Bajaj S, Hoff SB, Dougherty KG. Percutaneous cardiopulmonary bypass-supported coronary angioplasty in patients with unstable angina pectoris or myocardial infarction and a left ventricular ejection fraction < or = 25%. Am J Cardiol. 1996 Jan 1;77(1):14-9. doi: 10.1016/s0002-9149(97)89127-8. PMID 8540450
- [Result] Van Belle E, Blouard P, McFadden EP, Lablanche JM, Bauters C, Bertrand ME. Effects of stenting of recent or chronic coronary occlusions on late vessel patency and left ventricular function. Am J Cardiol. 1997 Nov 1;80(9):1150-4. doi: 10.1016/s0002-9149(97)00631-0. PMID 9359541
- [Result] Bax JJ, Poldermans D, Elhendy A, Cornel JH, Boersma E, Rambaldi R, Roelandt JR, Fioretti PM. Improvement of left ventricular ejection fraction, heart failure symptoms and prognosis after revascularization in patients with chronic coronary artery disease and viable myocardium detected by dobutamine stress echocardiography. J Am Coll Cardiol. 1999 Jul;34(1):163-9. doi: 10.1016/s0735-1097(99)00157-6. PMID 10400006